CLINICAL TRIAL: NCT00006392
Title: Selenium and Vitamin E Cancer Prevention Trial (SELECT) for Prostate Cancer
Brief Title: S0000 Selenium and Vitamin E in Preventing Prostate Cancer
Acronym: SELECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); Cancer and Leukemia Group B (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDR0000068277; S0000 (Other: SWOG); U10CA037429 (NIH); NCT00076128 (obsolete NCT alias)
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Results first posted 2012-11-06 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Vitamin E; alpha-Tocopherol; Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin E + selenium placebo (Experimental): vitamin E and selenium placebo daily for 7-12 years
  Interventions: Drug: Vitamin E; Other: selenium placebo
- Selenium + vitamin E placebo (Experimental): selenium and vitamin E placebo daily for 7-12 years
  Interventions: Drug: Selenium; Other: Vitamin E placebo
- Vitamin E + selenium (Experimental): vitamin E and selenium placebo daily for 7-12 years
  Interventions: Drug: Vitamin E; Drug: Selenium
- Vitamin E placebo + selenium placebo (Placebo Comparator): vitamine E placebo and selenium placebo daily for 7-12 years
  Interventions: Other: Vitamin E placebo; Other: selenium placebo

INTERVENTIONS:
Drug: Vitamin E — 400 IU daily by mouth for 7-12 years
  Other Names: alpha tocopherol
  Arms: Vitamin E + selenium; Vitamin E + selenium placebo
Drug: Selenium — 200 mcg daily for 7-12 years
  Other Names: L-selenomethionine
  Arms: Selenium + vitamin E placebo; Vitamin E + selenium
Other: Vitamin E placebo — daily for 7-12 years
  Other Names: placebo
  Arms: Selenium + vitamin E placebo; Vitamin E placebo + selenium placebo
Other: selenium placebo — daily for 7-12 years
  Other Names: placebo
  Arms: Vitamin E + selenium placebo; Vitamin E placebo + selenium placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. It is not yet known which regimen of selenium and/or vitamin E may be more effective in preventing prostate cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of selenium and vitamin E, either alone or together, in preventing prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of selenium and vitamin E administered alone vs in combination on the clinical incidence of prostate cancer.
* Compare the effect of these prevention regimens on the incidence of lung cancer, colorectal cancer, and all cancers combined in participants on this study.
* Compare the effect of these prevention regimens on prostate cancer-free survival, lung cancer-free survival, colorectal cancer-free survival, cancer-free survival, overall survival, and serious cardiovascular events in these participants.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy male volunteers
* Digital rectal examination (DRE) deemed not suspicious for prostate cancer performed within 364 days prior to study entry

  * Participants with a suspicious DRE are ineligible even if a recent or subsequent biopsy is negative for cancer
* Total prostate-specific antigen ≤ 4.0 ng/mL within 364 days prior to study entry
* No prior prostate cancer or high-grade (grade 2-3) prostatic intraepithelial neoplasia

PATIENT CHARACTERISTICS:

Age:

* See Disease Characteristics

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* Systolic blood pressure < 160 mm Hg
* Diastolic blood pressure < 90 mm Hg
* No history of hemorrhagic stroke

Other:

* No malignancies within the past 5 years except basal cell or squamous cell skin cancer
* No uncontrolled medical illness
* No retinitis pigmentosa

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 7 years since prior randomization to SWOG-9217, with completion of end-of-study biopsy requirement
* No additional concurrent selenium or vitamin E (contained in individual supplements, antioxidant mix, or multivitamin)
* Concurrent multivitamins allowed (supplied on study)
* No concurrent anticoagulation therapy (e.g., warfarin)
* Concurrent prophylactic aspirin (average daily dose no greater than 175 mg/day) allowed

  * Concurrent daily aspirin dose ≤ 81 mg for participants receiving clopidogrel
* Concurrent anti-hypertension medication allowed
* No concurrent participation in another study involving a medical, surgical, nutritional, or life-style intervention (unless no longer receiving the intervention and are in the follow-up phase only)

Ages: 50 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35533 (Actual)
Dates: Start 2001-07; Primary Completion 2011-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Klein, MD, Study Chair — The Cleveland Clinic; Philip J. Walther, MD, PhD, Study Chair — Duke University; Laurence H. Klotz, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre; Scott M. Lippman, M.D., Study Chair — MD Anderson; Ian M. Thompson, M.D., Study Chair — University of Texas; J. Michael Gaziano, M.D., Study Chair — MAVERIC; Daniel D Karp, M.D., Study Chair — Beth Israel Deaconess; Fadlo R. Khuri, M.D., Study Chair — MD Anderson; Michael M Lieber, M.D., Study Chair — Mayo Clinic
Locations (13):
- United States (13):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Good Samaritan Hospital Cancer Treatment Center, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - LaFortune Cancer Center at St. John Medical Center, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - U.T. Cancer Institute at University of Tennessee Medical Center, Knoxville, Tennessee

REFERENCES:
- [Background] Hoque A, Albanes D, Lippman SM, Spitz MR, Taylor PR, Klein EA, Thompson IM, Goodman P, Stanford JL, Crowley JJ, Coltman CA, Santella RM. Molecular epidemiologic studies within the Selenium and Vitamin E Cancer Prevention Trial (SELECT). Cancer Causes Control. 2001 Sep;12(7):627-33. doi: 10.1023/a:1011277600059. PMID 11552710
- [Background] El-Bayoumy K. The negative results of the SELECT study do not necessarily discredit the selenium-cancer prevention hypothesis. Nutr Cancer. 2009;61(3):285-6. doi: 10.1080/01635580902892829. No abstract available. PMID 19373601
- [Background] Cook ED, Moody-Thomas S, Anderson KB, Campbell R, Hamilton SJ, Harrington JM, Lippman SM, Minasian LM, Paskett ED, Craine S, Arnold KB, Probstfield JL. Minority recruitment to the Selenium and Vitamin E Cancer Prevention Trial (SELECT). Clin Trials. 2005;2(5):436-42. doi: 10.1191/1740774505cn111oa. PMID 16315648
- [Background] Kristal AR, King IB, Albanes D, Pollak MN, Stanzyk FZ, Santella RM, Hoque A. Centralized blood processing for the selenium and vitamin E cancer prevention trial: effects of delayed processing on carotenoids, tocopherols, insulin-like growth factor-I, insulin-like growth factor binding protein 3, steroid hormones, and lymphocyte viability. Cancer Epidemiol Biomarkers Prev. 2005 Mar;14(3):727-30. doi: 10.1158/1055-9965.EPI-04-0596. PMID 15767358
- [Background] Lippman SM, Goodman PJ, Klein EA, Parnes HL, Thompson IM Jr, Kristal AR, Santella RM, Probstfield JL, Moinpour CM, Albanes D, Taylor PR, Minasian LM, Hoque A, Thomas SM, Crowley JJ, Gaziano JM, Stanford JL, Cook ED, Fleshner NE, Lieber MM, Walther PJ, Khuri FR, Karp DD, Schwartz GG, Ford LG, Coltman CA Jr. Designing the Selenium and Vitamin E Cancer Prevention Trial (SELECT). J Natl Cancer Inst. 2005 Jan 19;97(2):94-102. doi: 10.1093/jnci/dji009. PMID 15657339
- [Result] Lippman SM, Klein EA, Goodman PJ, Lucia MS, Thompson IM, Ford LG, Parnes HL, Minasian LM, Gaziano JM, Hartline JA, Parsons JK, Bearden JD 3rd, Crawford ED, Goodman GE, Claudio J, Winquist E, Cook ED, Karp DD, Walther P, Lieber MM, Kristal AR, Darke AK, Arnold KB, Ganz PA, Santella RM, Albanes D, Taylor PR, Probstfield JL, Jagpal TJ, Crowley JJ, Meyskens FL Jr, Baker LH, Coltman CA Jr. Effect of selenium and vitamin E on risk of prostate cancer and other cancers: the Selenium and Vitamin E Cancer Prevention Trial (SELECT). JAMA. 2009 Jan 7;301(1):39-51. doi: 10.1001/jama.2008.864. Epub 2008 Dec 9. PMID 19066370
- [Result] Klein EA, Thompson IM Jr, Tangen CM, Crowley JJ, Lucia MS, Goodman PJ, Minasian LM, Ford LG, Parnes HL, Gaziano JM, Karp DD, Lieber MM, Walther PJ, Klotz L, Parsons JK, Chin JL, Darke AK, Lippman SM, Goodman GE, Meyskens FL Jr, Baker LH. Vitamin E and the risk of prostate cancer: the Selenium and Vitamin E Cancer Prevention Trial (SELECT). JAMA. 2011 Oct 12;306(14):1549-56. doi: 10.1001/jama.2011.1437. PMID 21990298
- [Derived] Tangen CM, Goodman PJ, Till C, Schenk JM, Lucia MS, Thompson IM Jr. Biases in Recommendations for and Acceptance of Prostate Biopsy Significantly Affect Assessment of Prostate Cancer Risk Factors: Results From Two Large Randomized Clinical Trials. J Clin Oncol. 2016 Dec 20;34(36):4338-4344. doi: 10.1200/JCO.2016.68.1965. Epub 2016 Oct 28. PMID 27998216
- [Derived] Goodman PJ, Tangen CM, Darke AK, Arnold KB, Hartline J, Yee M, Anderson K, Caban-Holt A, Christen WG, Cassano PA, Lance P, Klein EA, Crowley JJ, Minasian LM, Meyskens FL. Opportunities and challenges in incorporating ancillary studies into a cancer prevention randomized clinical trial. Trials. 2016 Aug 12;17:400. doi: 10.1186/s13063-016-1524-9. PMID 27519183
- [Derived] Chan JM, Darke AK, Penney KL, Tangen CM, Goodman PJ, Lee GM, Sun T, Peisch S, Tinianow AM, Rae JM, Klein EA, Thompson IM Jr, Kantoff PW, Mucci LA. Selenium- or Vitamin E-Related Gene Variants, Interaction with Supplementation, and Risk of High-Grade Prostate Cancer in SELECT. Cancer Epidemiol Biomarkers Prev. 2016 Jul;25(7):1050-1058. doi: 10.1158/1055-9965.EPI-16-0104. Epub 2016 May 6. PMID 27197287
- [Derived] Abner EL, Dennis BC, Mathews MJ, Mendiondo MS, Caban-Holt A, Kryscio RJ, Schmitt FA; PREADViSE Investigators; Crowley JJ; SELECT Investigators. Practice effects in a longitudinal, multi-center Alzheimer's disease prevention clinical trial. Trials. 2012 Nov 20;13:217. doi: 10.1186/1745-6215-13-217. PMID 23171483
- [Derived] Goodman PJ, Hartline JA, Tangen CM, Crowley JJ, Minasian LM, Klein EA, Cook ED, Darke AK, Arnold KB, Anderson K, Yee M, Meyskens FL, Baker LH. Moving a randomized clinical trial into an observational cohort. Clin Trials. 2013 Feb;10(1):131-42. doi: 10.1177/1740774512460345. Epub 2012 Oct 12. PMID 23064404
- [Derived] Chlebowski RT, Menon R, Chaisanguanthum RM, Jackson DM. Prospective evaluation of two recruitment strategies for a randomized controlled cancer prevention trial. Clin Trials. 2010 Dec;7(6):744-8. doi: 10.1177/1740774510383886. Epub 2010 Sep 10. PMID 20833684
- [Derived] Cook ED, Arnold KB, Hermos JA, McCaskill-Stevens W, Moody-Thomas S, Probstfield JL, Hamilton SJ, Campbell RD, Anderson KB, Minasian LM. Impact of supplemental site grants to increase African American accrual for the Selenium and Vitamin E Cancer Prevention Trial. Clin Trials. 2010 Feb;7(1):90-9. doi: 10.1177/1740774509357227. PMID 20156960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men were randomized at 427 study sites in the US, Puerto Rico and Canada between August 22, 2001 and June 24, 2004.
Pre-assignment Details: Prior to randomization, there was a three month formal pre-randomization period with no placebo run-in capsules to give potential participants to decide if they would agree to stop disallowed over-the-counter supplements of selenium or vitamin E. By returning for randomization, they exhibited their willingness to adhere to the trial.
Groups:
- Vitamin E: Vitamin E + matching placebo for selenium
- Selenium: Selenium + matching placebo for vitamin E
- Combination: Vitamin E + selenium
- Placebo: Matching placebo for vitamin E + matching placebo for selenium
Period: Overall Study
Arm/Group | Vitamin E | Selenium | Combination | Placebo
Started | 8904 | 8910 | 8863 | 8856
Completed | 8737 | 8752 | 8703 | 8696
Not Completed | 167 | 158 | 160 | 160
Not completed — Ineligible | 11 | 3 | 5 | 5
Not completed — Poor data/ppt mgmt, regulatory problems | 156 | 155 | 155 | 155

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin E | Selenium | Combination | Placebo | Total
Number analyzed (Participants) | 8737 | 8752 | 8703 | 8696 | 34888
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.4 [58.1 to 67.8] | 62.6 [58.1 to 67.8] | 62.3 [58.0 to 67.8] | 62.6 [58.2 to 68.0] | 62.3 [58.1 to 67.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 8737 | 8752 | 8703 | 8696 | 34888
Race/Ethnicity, Customized [Number; unit: Participant]
  White | 6890 | 6942 | 6874 | 6863 | 27569
  African American | 1107 | 1053 | 1076 | 1078 | 4314
  Hispanic (non-African American) | 477 | 481 | 484 | 492 | 1934
  Hispanic (African American) | 103 | 86 | 95 | 76 | 360
  Other | 160 | 190 | 174 | 187 | 711
Region of Enrollment [Number; unit: participants]
  United States | 7463 | 7471 | 7427 | 7428 | 29789
  Canada | 909 | 915 | 911 | 904 | 3639
  Puerto Rico | 365 | 366 | 365 | 364 | 1460
Age (categorical) [Number; unit: participants]
  50 - 54 years | 402 | 337 | 385 | 355 | 1479
  55 - 64 years | 5143 | 5076 | 5052 | 5078 | 20349
  65 - 74 years | 2641 | 2733 | 2731 | 2702 | 10807
  >= 75 years | 551 | 606 | 535 | 561 | 2253
Education (highest) [Number; unit: Participant]
  <= High school graduate or GED | 1875 | 1917 | 1898 | 1993 | 7683
  Some college/vocational school | 2387 | 2327 | 2348 | 2291 | 9353
  >= College graduate | 4394 | 4430 | 4372 | 4317 | 17513
  Unknown/missing | 81 | 78 | 85 | 95 | 339
PSA (ng/ml) [Number; unit: Participant]
  0.1 - 1.0 | 4208 | 4218 | 4213 | 4122 | 16761
  1.1 - 2.0 | 2653 | 2661 | 2666 | 2728 | 10708
  2.1 - 3.0 | 1228 | 1211 | 1149 | 1168 | 4756
  3.1 - 4.0 | 634 | 652 | 659 | 666 | 2611
  > 4.0 | 3 | 2 | 1 | 5 | 11
  Unknown/missing | 11 | 8 | 15 | 7 | 41
Smoking status [Number; unit: Participant]
  Never | 3752 | 3780 | 3666 | 3682 | 14880
  Current | 659 | 631 | 670 | 655 | 2615
  Former | 4194 | 4214 | 4242 | 4208 | 16858
  Ever (unknown status) | 55 | 61 | 56 | 63 | 235
  Unknown | 77 | 66 | 69 | 88 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prostate Cancer
Description: Participants are seen at the study site every six month for an update of medical events. Prostate cancer diagnosis is based on participant report followed by the submission of a pathologic sample to central pathology review for confirmation.
Time Frame: Every six months for 7 to 12 years depending on when the participant was randomized.
Population: All randomized eligible men not at 2 sites for which the DSMC said the data could not be used due to participant and data management issues as well as regulatory problems.
Measure: Number; unit: participants
Arm/Group | Vitamin E | Selenium | Combination | Placebo
Number analyzed (Participants) | 8737 | 8752 | 8703 | 8696
participants | 473 | 432 | 437 | 416
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Per study design, with a sample size of 32,400 men, using a 1-sided alpha=.005 level (equivalent to a 2-sided alpha=.01 level) there was 96% power to detect a 25% reduction in prostate cancer for either agent vs. Placebo; Test type: Superiority or Other; p < .01, Regression, Cox — The p-value was adjusted for multiple comparisons; Hazard Ratio (HR) = 1.13, 99% CI 2-sided [0.95 to 1.35]
Statistical Analysis 2: Comparison: Selenium vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .01, Regression, Cox — The p-value was adjusted for multiple comparisons; Hazard Ratio (HR) = 1.04, 99% CI 2-sided [0.87 to 1.24]
Statistical Analysis 3: Comparison: Combination vs Placebo; Per study design, with a sample size of 32,400 men, using a 1-sided alpha=.005 level (equivalent to a 2-sided alpha=.01 level) there was 99% power to detect a 44% reduction in prostate cancer for combination vs. Placebo; Test type: Superiority or Other; p < .01, Regression, Cox — The p-value was adjusted for multiple comparisons; Hazard Ratio (HR) = 1.05, 99% CI [.88 to 1.25]

2. Secondary Outcome: Number of Participants With Lung Cancer
Description: Participants are seen at the study site every six month for an update of medical events. Cancer diagnoses are based on participant report. Medical records for non-prostate cancers were collected but they were not pathologically confirmed. If the participant has been diagnosed with prostate cancer, study site visits are once a year. Follow-up was planned for seven to 12 years depending on when the participant was randomized.
Time Frame: Participants are assessed for medical every six months for 7 to 12 years depending on when he was randomized . Upon diagnosis of prostate cancer, updates are annual.
Population: All randomized eligible participants excluding all men from 2 study sites that the DSMC said to exclude due to poor participant/data management and regulatory issues.
Measure: Number; unit: participants
Arm/Group | Vitamin E | Selenium | Combination | Placebo
Number analyzed (Participants) | 8737 | 8752 | 8703 | 8696
participants | 67 | 75 | 78 | 67
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p > .05, Regression, Cox — The trial was designed to study prostate cancer and lung cancer has a lower incidence rate, there was limited power to look at lung cancer incidence. A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Hazard Ratio (HR) = 1.0, 99% CI [.64 to 1.55] — The placebo was the denominator
Statistical Analysis 2: Comparison: Selenium vs Placebo; Test type: Superiority or Other; p > .01, Regression, Cox — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.12, 99% CI 2-sided [0.73 to 1.72] — The placebo was the denominator
Statistical Analysis 3: Comparison: Combination vs Placebo; Test type: Superiority or Other; p > .01, Regression, Cox — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.16, 99% CI 2-sided [0.90 to 1.16] — The placebo was the denominator

3. Secondary Outcome: Number of Participants With Colorectal Cancer
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Vitamin E | Selenium | Combination | Placebo
Number analyzed (Participants) | 8737 | 8752 | 8703 | 8696
participants | 66 | 63 | 77 | 60
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; The trial was designed to study prostate cancer and colorectal cancer has a lower incidence rate, there was limited power to look at colorectal cancer incidence; Test type: Superiority or Other; p > .05, Regression, Cox — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Hazard Ratio (HR) = 1.09, 99% CI 2-sided [0.69 to 1.73] — The placebo was the denominator
Statistical Analysis 2: Comparison: Selenium vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p > .05, Regression, Cox — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Hazard Ratio (HR) = 1.05, 99% CI 2-sided [0.66 to 1.67] — The placebo was the denominator
Statistical Analysis 3: Comparison: Combination vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p > .05, Regression, Cox — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Hazard Ratio (HR) = 1.28, 99% CI 2-sided [0.82 to 2.00] — The placebo was the denominator

4. Secondary Outcome: Number of Participants With Any Diagnosis of Cancer
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Vitamin E | Selenium | Combination | Placebo
Number analyzed (Participants) | 8737 | 8752 | 8703 | 8696
participants | 856 | 837 | 846 | 824
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; The power to look at all cancer incidence is greater than 90%; Test type: Superiority or Other; p > .05, Regression, Cox — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Hazard Ratio (HR) = 1.03, 99% CI 2-sided [0.91 to 1.17] — The placebo was the denominator
Statistical Analysis 2: Comparison: Selenium vs Placebo; The power to look at all cancer incidence is greater than 90%; Test type: Superiority or Other; p > .05, Regression, Cox — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Hazard Ratio (HR) = 1.01, 99% CI 2-sided [0.89 to 1.15] — The placebo was the denominator
Statistical Analysis 3: Comparison: Combination vs Placebo; The power to look at all cancer incidence is greater than 90%; Test type: Superiority or Other; p > .05, Regression, Cox — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Hazard Ratio (HR) = 1.02, 99% CI [0.90 to 1.16] — The placebo was the denominator

5. Secondary Outcome: Prostate Cancer Free Survival; Lung Cancer-free Survival, Colorectal Cancer-free Survival, Cancer-free Survival, Overall Survival
Description: Participants are seen at the study site every six month for an update of medical events. If the participant has been diagnosed with prostate cancer, study site visits are once a year. Prostate cancer diagnosis is based on participant report followed by the submission of a pathologic sample to central pathology review for confirmation. Other cancer diagnoses are based on participant report. Medical records for non-prostate cancers were collected but they were not pathologically confirmed. Follow-up was planned for seven to 12 years depending on when the participant was randomized.
Time Frame: as for outcome 2
Population: All randomized eligible participants excluding all men from 2 study sites that the DSMC said to exclude due to poor participant/data management and regulatory issues. Deaths include those reported as SAEs as well as non-SAE deaths as this was a prevention trial with older generally healthy men at baseline who were followed for a long time.
Measure: Number; unit: participants
Arm/Group | Vitamin E | Selenium | Combination | Placebo
Number analyzed (Participants) | 8737 | 8752 | 8703 | 8696
participants
  All deaths | 358 | 378 | 359 | 382
  All cancer deaths | 106 | 128 | 117 | 125
  Prostate cancer deaths | 0 | 1 | 0 | 0
  Lung cancer deaths | 38 | 45 | 39 | 41
  Colorectal cancer deaths | 13 | 10 | 15 | 10
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Only results from overall survival are presented as the number of cancer-specific deaths is too few to be meaningful; Test type: Superiority or Other; p > .05, Regression, Cox — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Hazard Ratio (HR) = 0.93, 99% CI [0.77 to 1.13] — The placebo is the denominator
Statistical Analysis 2: Comparison: Selenium vs Placebo; Only results from overall survival are presented as the number of cancer-specific deaths is too few to be meaningful; Test type: Superiority or Other; p > .05, Regression, Cox — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Hazard Ratio (HR) = 0.99, 99% CI 2-sided [0.82 to 1.19] — The placebo was the denominator
Statistical Analysis 3: Comparison: Combination vs Placebo; Only results from overall survival are presented as the number of cancer-specific deaths is too few to be meaningful; Test type: Superiority or Other; p > .05, Regression, Cox — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Hazard Ratio (HR) = 0.94, 99% CI 2-sided [0.77 to 1.13]

6. Secondary Outcome: Number of Participants With Serious Cardiovascular Events
Description: Participants are seen at the study site every six month for an update of medical events. If the participant has been diagnosed with prostate cancer, study site visits are once a year. Cardiovascular events are based on self-report and are not confirmed. Follow-up was planned for seven to 12 years depending on when the participant was randomized.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Vitamin E | Selenium | Combination | Placebo
Number analyzed (Participants) | 8737 | 8752 | 8703 | 8696
participants | 1034 | 1080 | 1041 | 1050
Statistical Analysis 1: Comparison: Vitamin E vs Placebo; Test type: Superiority or Other; p > .05, Chi-squared — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Risk Ratio (RR) = 0.98, 99% CI 2-sided [0.88 to 1.09] — The placebo was the denominator
Statistical Analysis 2: Comparison: Selenium vs Placebo; Test type: Superiority or Other; p > .05, Chi-squared — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Risk Ratio (RR) = 1.02, 99% CI 2-sided [0.92 to 1.13] — The placebo was the denominator
Statistical Analysis 3: Comparison: Combination vs Placebo; Test type: Superiority or Other; p > .05, Chi-squared — A 99% CI (rather than a 95% CI) was used to adjust for the multiple comparisons; Risk Ratio (RR) = 0.99, 99% CI 2-sided [0.89 to 1.10] — The placebo was the denominator

ADVERSE EVENTS:
Time Frame: 6 months
Description: Study site visits, collected by CRA based on participant interview and annual limited physical exam
Groups:
- Selenium Alone: Selenium + placebo for vitamin E
- Combination: Selenium + vitamin E
- Placebo: Placebo for selenium + placebo for vitamin E
- Vitamin E Alone: Vitamin E + placebo for selenium
Arm/Group | Selenium Alone | Combination | Placebo | Vitamin E Alone
Serious Adverse Events (participants affected / at risk) | 96/8752 | 93/8702 | 108/8696 | 99/8737
Other Adverse Events (participants affected / at risk) | 2605/8752 | 2550/8702 | 2421/8696 | 2553/8737
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selenium Alone (N=8752) | Combination (N=8702) | Placebo (N=8696) | Vitamin E Alone (N=8737)
Arrhythmia, NOS (Cardiac disorders) | 3 | 2 | 1 | 0
Cardiac ischemia/infarction (Cardiac disorders) | 25 | 26 | 27 | 18
Cardiovascular-other (Cardiac disorders) | 9 | 12 | 17 | 14
Conduction abnormality/block (Cardiac disorders) | 0 | 1 | 1 | 0
LVEF decrease/CHF (Cardiac disorders) | 9 | 2 | 1 | 4
Supraventricular arrhythmia (Cardiac disorders) | 3 | 0 | 3 | 1
Ventricular arrhythmia (Cardiac disorders) | 2 | 2 | 8 | 3
Eye-other (Eye disorders) | 0 | 0 | 0 | 1
Vision,NOS (Eye disorders) | 0 | 0 | 1 | 0
Dyspepsia/heartburn (Gastrointestinal disorders) | 0 | 0 | 1 | 0
GI-other (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Melena/ GI bleeding (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Constitutional symptoms-other (General disorders) | 0 | 0 | 1 | 0
Hemorrhage w/o 3-4 thrombocyt (General disorders) | 0 | 0 | 0 | 1
Pain-other (General disorders) | 1 | 0 | 0 | 0
Reportable adverse event, NOS (General disorders) | 11 | 10 | 17 | 19
Liver-clinical (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Liver-other (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Respiratory infect w/o neutrop (Infections and infestations) | 2 | 1 | 1 | 1
Respiratory infection, unk ANC (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tr infect w/o neutrop (Infections and infestations) | 0 | 1 | 0 | 0
Surgery-hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Weight gain (Investigations) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia/arthralgia, NOS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Second primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 2 | 3
CNS hemorrhage (Nervous system disorders) | 8 | 8 | 3 | 9
Cerebrovascular ischemia (Nervous system disorders) | 7 | 17 | 10 | 8
Cranial neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Neuro-other (Nervous system disorders) | 1 | 0 | 2 | 0
Seizures (Nervous system disorders) | 1 | 0 | 0 | 0
Sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Erectile impotence (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Emphysema/COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Aortic Stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Cardiomyopathy (Vascular disorders) | 0 | 0 | 0 | 1
Carotid stenosis (Vascular disorders) | 0 | 2 | 0 | 2
Hypertension (Vascular disorders) | 2 | 1 | 0 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral arterial ischemia (Vascular disorders) | 1 | 1 | 1 | 1
Thrombosis/embolism (Vascular disorders) | 2 | 2 | 3 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selenium Alone (N=8752) | Combination (N=8702) | Placebo (N=8696) | Vitamin E Alone (N=8737)
Cardiac ischemia/infarction (Cardiac disorders) | 558 | 533 | 529 | 551
Halitosis (Gastrointestinal disorders) | 523 | 555 | 447 | 517
Fatigue/malaise/lethargy (General disorders) | 698 | 657 | 632 | 660
Dermatitis (Skin and subcutaneous tissue disorders) | 647 | 593 | 554 | 627
Nail changes (Skin and subcutaneous tissue disorders) | 1129 | 1080 | 1072 | 1070

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No